CLINICAL TRIAL: NCT03023371
Title: National Registry of IgG4-RD in China
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Other Study IDs: IgG4-RD Group in China
Record Dates: First submitted 2017-01-02; First posted 2017-01-18 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: IgG4-Related Disease
Keywords: Registry; cohort study; IgG4-related disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Peripheral blood samples from IgG4-RD patients will be saved for DNA extration and study.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to establish a nation-wide cohort study of IgG4-related disease (IgG4-RD) in China.

Methods: All the patients fulfilling diagnostic criteria of IgG4-RD (2011) would be enrolled from multi-centers around China. A online database system has been established.

Endpoints: The primary endpoint is to investigate the clinical manifestations of Chinese IgG4-RD patients; the secondary endpoints including the demographic features,laboratory characteristics, immunological tests, imaging and pathological features, in addition, the treatment and prognosis of the disease.

DETAILED DESCRIPTION:
This is a multicenter registry study of IgG4-RD patients. Newly diagnosed IgG4-RD patients will be recruited from allover the China. Inclusion criteria: patients with definite, probable, or possible IgG4-RD according to the 2011 comprehensive diagnostic criteria for IgG4-RD will be recruited. Exclusion criteria: patients with malignancy or other autoimmune diseases are excluded.

The data will be uploaded through the platform of Chinese Rheumatology Information Platform. Demographic data, initial symptoms, disease duration, history of allergy, and physical examination, organ involvements, laboratory findings, radiological and pathological results, as well as treatment, side effects will be recorded.

This study was approved by the Medical Ethics Committee of PUMCH (Beijing, China). All patients will signe informed consent.

Statistical Analysis: All parameters are described in the standard summary statistics, including mean, standard deviation, minimum, and maximum. All statistical analyses will be performed by SPSS.

Endpoints: The primary endpoint is to investigate the organ involvements of Chinese IgG4-RD patients. The secondary endpoints including the demographic features,laboratory characteristics, immunological tests, imaging and pathological features, in addition, the treatment and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Conforming to the diagnostic criteria of IgG4-RD (2011);

Exclusion Criteria:

* Excluding other mimicing IgG4-RD, including tumors, vasculitis and sarcoidosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IgG4-RD patients around China
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Organ involvements of Chinese IgG4-RD patients | 5 years
  To calculate the percentage of organ involvements in at least 900 patients.

SECONDARY OUTCOMES:
Response rate of glucocorticoids and immunosuppressants on IgG4-RD in China | 5 years
Relapse rate of IgG4-RD patients in China | 5 years
The correlation between baseline disease activities and relapse rate. | 5 years
The incidence rate of tumor in IgG4 related disease patients in China. | 5 years
Ten year survival rate of patients with IgG4 related disease in China. | 10 years
The imaging features of involved organs. | 3 years
The sensitivity and specificity of IgG4 positive plasma cells in pathological diagnosis of IgG4 related disease. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes